CLINICAL TRIAL: NCT00023647
Title: A Phase I Dose-Ranging Safety Study Using Intranodal Delivery of a Plasmid DNA (Synchrotope TA2M) in Adult Stage IV Melanoma Patients
Brief Title: Vaccine Therapy in Treating Patients With Stage IV Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068847; CTL-207-216; CTL-BB-IND-9146; LAC-USC-10M001; NCI-V01-1666
Record Dates: First submitted 2001-09-13; First posted 2004-02-16 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Synchrotope TA2M, 800 micrograms (Experimental): Tyrosinase peptides, 800 micrograms
  Interventions: Biological: Synchrotope TA2M
- Synchrotope TA2M, 200 micrograms (Experimental): Tyrosinase peptides, 200 micrograms
  Interventions: Biological: Synchrotope TA2M
- Synchrotope TA2M, 400 micrograms (Experimental): Tyrosinase peptides, 400 micrograms
  Interventions: Biological: Synchrotope TA2M

INTERVENTIONS:
Biological: Synchrotope TA2M — Cancer Vaccine, Immunotherapy
  Arms: Synchrotope TA2M, 800 micrograms
Biological: Synchrotope TA2M — Cancer Vaccine, Immunotherapy
  Arms: Synchrotope TA2M, 200 micrograms
Biological: Synchrotope TA2M — Cancer Vaccine, Immunotherapy
  Arms: Synchrotope TA2M, 400 micrograms

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells. Infusing the vaccine directly into a lymph node may cause a stronger immune response and kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of vaccine therapy given directly into a lymph node in treating patients who have stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety and tolerability of intranodal Synchrotope TA2M plasmid DNA vaccine in patients with stage IV melanoma. II. Determine the immune response of patients treated with this vaccine. III. Determine the clinical response of patients treated with this vaccine.

OUTLINE: This is dose-escalation, multicenter study. Patients receive Synchrotope TA2M plasmid DNA vaccine intranodally continuously over 96 hours beginning on days 0, 14, 28, and 42. Treatment continues for up to 2 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 8 patients receive escalating doses of Synchrotope TA2M plasmid DNA vaccine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which no more than 2 of 8 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: Approximately 16-24 patients will be accrued for this study within 12 months.

ELIGIBILITY:
INCLUSION CRITERIA - Patient must meet the following during the screening and baseline visits:

1. The patients or their legally acceptable representative must give signed informed consent for participation in the study before any study procedure is performed.
2. Patients must be 18 years of age or older at pre-study
3. Patients must be ambulatory, ECOG performance status of 0 or 1 (Appendix II)
4. Patients have histologically confirmed diagnosis of Stage IV melanoma according to AJCC/UICC modified system with an expected survival time of more than 3 months
5. Patients must be positive for HLA-A2 (Patients tested positive within 5 years of pre-study screening do not need to be tested again for HLA-A2)
6. Patients must agree to use an acceptable method of birth control

   1. intrauterine device
   2. oral hormonal contraception
   3. combination of spermicide and barrier method or
   4. abstinence
7. Female patients of childbearing potential must have a confirmed negative urine pregnancy test on Day 0

EXCLUSION CRITERIA - Patients meeting any of the following criteria will NOT be eligible for the study:

1. Patients who have hematological abnormalities as evidenced by:

   1. Neutrophils < 1,500/mm3
   2. Leukocytes < 3,000/mm3
   3. Platelets < 75,000/mm3
   4. Hemoglobin < 9.0 g/dL
2. Patients who have hepatic disease as evidenced by:

   1. SGOT/SGPT (AST/ALT) > 2.5 x the upper limit of normal (ULN)
   2. alkaline phosphatase > 2.5 x ULN
   3. Bilirubin > 1.5 x ULN\
   4. positive for hepatitis B surface antigen
   5. positive for hepatitis C antibody
3. Patients who have known or suspected renal impairment as evidenced by:

   1. serum creatinine > 1.5 x ULN, and/or
   2. serum urea > 2.6 x ULN
4. Patients with a history of ocular melanoma
5. Patients with brain metastases, unless completed resected
6. Patients with a positive HIV antibody test
7. Patients with medical, sociological, or psychological impediments that may compromise compliance with the protocol
8. Patients who are nursing, pregnant or planning to become pregnant within 6 months of treatment completion
9. Patients who are receiving chemo-, radio- or immunotherapy concurrently or within the preceding four weeks
10. Patients who are taking drugs that affect immune function such as systemic corticosteroids or immunomodulatory drugs concurrently or within the preceding four weeks
11. Patients who are receiving any investigational drug concurrently or within the preceding four weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2000-07; Primary Completion 2002-04 (Actual); Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events assessed by complete blood count, blood chemistry, polymerase chain reaction, physical examination and urinalysis | Individual 96-hour infusion periods on days 0, 14, 28 and 42 and on day 56

SECONDARY OUTCOMES:
Change in magnitude of antigen-specific cytotoxic t-lymphocyte in peripheral blood mononuclear cells | Day 0 (pre-study), last day of individual 96-hour infusion periods (days 4, 17, 31 and 45) and on day 56
Assessment of delayed-type hypersensitivity to intradermal injections 24 hours after injection | Days 1, 29 and 57
Change in size of target lesions by x-ray computed tomography before (day 0) and after (day 56)treatment | Change from pre-study (day 0) to day 56

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Hickingbottom, JD, MD, Study Chair — Mannkind Corporation
Locations (1):
- USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California, United States

REFERENCES:
- [Result] Tagawa ST, Lee P, Snively J, Boswell W, Ounpraseuth S, Lee S, Hickingbottom B, Smith J, Johnson D, Weber JS. Phase I study of intranodal delivery of a plasmid DNA vaccine for patients with Stage IV melanoma. Cancer. 2003 Jul 1;98(1):144-54. doi: 10.1002/cncr.11462. PMID 12833467